CLINICAL TRIAL: NCT06642584
Title: A Study Investigating the Pharmacokinetic Properties When Dosing Different Formulations of Semaglutide to Healthy Male Participants
Brief Title: A Research Study Looking at New Protein-based Tablets in Healthy Men - Oral Formulation IV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9501-5006; U1111-1304-9627 (Other: World Health Organisation (WHO))
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers Type 2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1: Semaglutide J then Semaglutide L (Experimental): Participants will receive subcutaneously semagutide B in treatment period 1 followed by oral semaglutide J then semaglutide L in treatment period 2.
  Interventions: Drug: Semaglutide B; Drug: Semaglutide J; Drug: Semaglutide L
- Sequence 2: Semaglutide L then Semaglutide J (Experimental): Participants will receive subcutaneously semagutide B in treatment period 1 followed by oral semaglutide L then semaglutide J in treatment period 2.
  Interventions: Drug: Semaglutide B; Drug: Semaglutide J; Drug: Semaglutide L
- Sequence 3: Semaglutide J then Semaglutide M (Experimental): Participants will receive subcutaneously semagutide B in treatment period 1 followed by oral semaglutide J then semaglutide M in treatment period 2.
  Interventions: Drug: Semaglutide B; Drug: Semaglutide J; Drug: Semaglutide M
- Sequence 4: Semaglutide M then Semaglutide J (Experimental): Participants will receive subcutaneously semagutide B in treatment period 1 followed by oral semaglutide M then semaglutide J in treatment period 2.
  Interventions: Drug: Semaglutide B; Drug: Semaglutide J; Drug: Semaglutide M
- Sequence 5: Semaglutide J then Semaglutide N (Experimental): Participants will receive subcutaneously semagutide B in treatment period 1 followed by oral semaglutide J then semaglutide N in treatment period 2.
  Interventions: Drug: Semaglutide B; Drug: Semaglutide J; Drug: Semaglutide N
- Sequence 6: Semaglutide N then Semaglutide J (Experimental): Participants will receive subcutaneously semagutide B in treatment period 1 followed by oral semaglutide N then semaglutide J in treatment period 2.
  Interventions: Drug: Semaglutide B; Drug: Semaglutide J; Drug: Semaglutide N

INTERVENTIONS:
Drug: Semaglutide B — Semaglutide B will be administered subcutaneously.
Drug: Semaglutide J — Semaglutide J will be administered as oral tablets.
Drug: Semaglutide L — Semaglutide L will be administered as oral tablets.
  Arms: Sequence 1: Semaglutide J then Semaglutide L; Sequence 2: Semaglutide L then Semaglutide J
Drug: Semaglutide M — Semaglutide M will be administered as oral tablets.
  Arms: Sequence 3: Semaglutide J then Semaglutide M; Sequence 4: Semaglutide M then Semaglutide J
Drug: Semaglutide N — Semaglutide N will be administered as oral tablets.
  Arms: Sequence 5: Semaglutide J then Semaglutide N; Sequence 6: Semaglutide N then Semaglutide J

SUMMARY:
This study is conducted to compare four different tablets containing the investigational medicine semaglutide at the same dose. It is done to test how semaglutide in each of the tablet versions is taken up in the body. Which treatments participants will receive is decided by chance. The study will last for about 28 weeks. The study will enroll healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male.
2. Age 18-64 years (both inclusive) at the time of signing the informed consent.
3. Body mass index (BMI) between 22.0 and 31.9 kilogram per square meter (kg/m^2) (both inclusive) at screening.
4. Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

1. Known or suspected hypersensitivity to study interventions or related products.
2. Any condition which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
3. Use of prescription medicinal products or non-prescription drugs, except routine vitamins, topical medication not reaching the systemic circulation and occasional use of paracetamol (acetaminophen) and ibuprofen, within 14 days prior to first dosing.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Adjusted AUC(sema); adjusted area under the semaglutide plasma concentration-time curve | From 0 to 24 hours after dosing on Days 122 and 132.
  Measured in hours nanomoles per liter (h * nmol/L).
Adjusted Cmax,(sema); adjusted maximum observed semaglutide plasma concentration | From 0 to 24 hours after dosing on Days 122 and 132.
  Measured in nanomoles per liter(nmol/L).
Adjusted tmax,sema; time to adjusted maximum observed semaglutide plasma concentration | From 0 to 24 hours after dosing on Days 122 and 132.
  Measured in hours.
t½,sema; the terminal half-life of semaglutide | From 0 to 840 hours after dosing on Day 132.
  Measured in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: https://novonordisk-trials.com